CLINICAL TRIAL: NCT07039201
Title: An Exploratory Clinical Study on the Safety and Efficacy of Autologous Chimeric Antigen Receptor T Cells Targeting Glypican-3 (CG-102-12C) in the Treament of Advanced Hepatocellular Carcinoma
Brief Title: A Study to Evaluate CG-102-12C in Glypican-3 (GPC3) Positive Advanced Hepatocellular Carcinoma (HCC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Cells & Genes Biotech (Unknown)
Responsible Party: Principal Investigator, TingBo Liang, Director physician, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG-102-12C
Record Dates: First submitted 2025-03-22; First posted 2025-06-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
Keywords: Advanced Hepatocellular Carcinoma; Chimeric antigen receptor T Cell; GPC3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Biological: CG-102-12C

INTERVENTIONS:
Biological: CG-102-12C — Chimeric Antigen Receptor Autologous T-cell

SUMMARY:
This study is a single-centre, single-arm, open-label, dose-escalation exploratory study with single-dose administration. Its objective is to evaluate the safety, tolerability, dose, anti-tumor efficacy, and pharmacokinetic characteristics of CG-102-12C in the participants with GPC3-positive advanced hepatocellular carcinoma who previously received adequate but uneffective systemic standard treatments.

DETAILED DESCRIPTION:
This study is a single-centre, open-label, dose-escalation exploratory clinical trial. Its objective is to evaluate the safety, tolerability, recommended dose, anti-tumor efficacy, and pharmacokinetic characteristics of CG-102-12C infused in participants with GPC3-positive advanced hepatocellular carcinoma who previously received adequate systemic standard treatments. The study will be carried out in accordance with the protocol. Due to the early-stage of the exploratory clinical research,, the anticipated sample size for the three dose groups is 7-12 participants.

ELIGIBILITY:
Inclusion Criteria:

* 1. The study participant has fully understood the potential risks and benefits of participating in this study and has signed the informed consent form.
* 2. Aged 18-75 years (inclusive of 18 and 75 years old).
* 3. Patients with advanced hepatocellular carcinoma (HCC) confirmed by histopathological or cytological examination to be GPC3-positive (advanced HCC is defined as Barcelona Clinic Liver Cancer (BCLC) stage C or stage B that is unsuitable for or has progressed after local treatment, including ablation therapy, interventional therapy, and radiotherapy). Patients must have previously received systemic standard treatment and experienced treatment failure or intolerance (systemic treatments include, but are not limited to, chemotherapy and molecular targeted therapy). Treatment failure is defined as disease progression during or after the most recent treatment.
* 4. Immunohistochemical analysis of tumor tissue samples must show GPC3 positivity (defined as >25% of pathological specimens with IHC-detected GPC3-positive cells and staining intensity ≥1+). Preferably ,target lesion specimens will be used, including freshly obtained tumor pathology samples or archived tumor pathology samples deemed acceptable by the investigator.
* 5. Child-Pugh score ≤7.
* 6. At least one evaluable tumor lesion as assessed by RECIST 1.1.
* 7. ECOG performance status score of 0-2.
* 8. Expected survival ≥3 months.
* 9. Hematological parameters must meet the following criteria:Absolute neutrophil count (ANC) ≥1×10^9/L;Absolute lymphocyte count (ALC) ≥0.5×10^9/L;Platelets ≥50×10^9/L;Hemoglobin ≥60 g/L or hematocrit >0.24.(No treatment with hematopoietic growth factors or blood transfusion within 3 days prior to laboratory tests).
* 10.Blood biochemistry must meet the following criteria:Total bilirubin (TBIL) ≤2.5 times the upper limit of normal (ULN);AST and ALT ≤5.0 times ULN;Serum albumin ≥28 g/L;Serum creatinine ≤1.5 times ULN;Creatinine clearance >50 mL/min (calculated using the Cockcroft-Gault formula).
* 11.Coagulation parameters must meet the following criteria:INR <1.5 times ULN;APTT <1.5 times ULN;PT prolongation ≤4 seconds.
* 12.If the patient is HBsAg positive or HBcAb positive, it is required that HBV-DNA ≤2000 IU/mL;
* 13.At screening, during apheresis, and within 3 days prior to preconditioning, female study participants of childbearing potential must have a negative blood pregnancy test; during the study period and for at least 1 year after completion of the study treatment, study participants of childbearing potential and their partners must use effective contraception.

Exclusion Criteria:

* 1. History of a second primary malignancy is permitted, unless the patient has undergone potentially curative treatment and has been free of the disease for 5 years.

Note: This time requirement (i.e., within 5 years) does not apply to patients with adequately treated carcinoma in situ of the cervix, localized squamous cell carcinoma of the skin, basal cell carcinoma, localized prostate cancer, ductal carcinoma in situ of the breast, or urothelial carcinoma <T1. Patients with prostate cancer under active surveillance are also eligible, or patients deemed eligible by the investigator after thorough evaluation.

* 2. Prior treatment with CAR-T or TCR-T cell therapy targeting any antigen or therapeutic cancer vaccines; or prior treatment with any therapy targeting GPC3.
* 3. Prior to apheresis, the patient has received the following antitumor therapies: Cytotoxic therapy within 14 days; Small molecule targeted therapy, epigenetic therapy, or experimental drug therapy within 14 days or at least 5 half-lives (whichever is longer), or treatment with invasive experimental medical devices; Monoclonal antibody therapy within 21 days; Immunomodulatory therapy within 7 days; Radiotherapy within 14 days.
* 4. Toxicities from prior antitumor therapies have not recovered to ≤ Grade 1 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE version 5.0), except for alopecia, Grade 2 peripheral neuropathy, and hypothyroidism controlled by hormone replacement therapy.
* 5. History of organ transplantation or currently awaiting organ transplantation (including liver transplantation).
* 6. Brain metastases with central nervous system symptoms or other clinically significant central nervous system diseases.
* 7. History of hepatic encephalopathy or current presence of hepatic encephalopathy.
* 8. Ascites requiring therapeutic intervention (excluding any ascites detected by imaging that does not require clinical intervention).
* 9. HCC tumor volume occupying ≥50% of the normal liver volume based on imaging, or presence of tumor thrombus in the main portal vein or inferior vena cava, or patients deemed ineligible by the investigator.
* 10.Women who are pregnant or breastfeeding.
* 11.Positive screening for hepatitis C virus antibody (HCV-Ab) or human immunodeficiency virus antibody (HIV-Ab); active syphilis. (Patients with positive HCV antibody but HCV-RNA below the detection limit of the research center are allowed to enroll).
* 12.Presence of severe underlying diseases, such as: Evidence of severe active viral, bacterial, or uncontrolled systemic fungal infections; Active or unstable autoimmune diseases or a history of autoimmune diseases within the past 3 years with potential for recurrence (including, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism; patients with vitiligo; childhood asthma that has completely resolved and requires no intervention in adulthood may be included; asthma requiring medical intervention with bronchodilators is excluded); Uncontrolled diabetes; Severe congestive heart failure classified as New York Heart Association (NYHA) Class III or above, or patients with an ejection fraction <50%; history of myocardial infarction or unstable angina within 6 months prior to treatment; Hypertension that cannot be controlled to the following range (systolic blood pressure <160 mmHg, diastolic blood pressure <100 mmHg) despite treatment with two antihypertensive medications; Clinically significant ventricular arrhythmias, or a history of unexplained syncope not due to vasovagal causes or dehydration; patients with constrictive pericarditis, significant pericardial effusion, cardiomyopathy, low voltage on limb leads of electrocardiogram, or other cardiac conditions deemed unsuitable by the investigator; Patients with clinically significant dementia, altered mental status, or a history of poorly controlled psychiatric disorders.
* 13.History of stroke or seizure within 6 months prior to signing the ICF.
* 14.Significant bleeding tendency, such as active gastrointestinal bleeding or coagulation disorders.
* 15.Chronic diseases requiring systemic corticosteroids or other immunosuppressive therapy, or treatment with systemic corticosteroids (≥70 mg prednisone or equivalent doses of other corticosteroids) or other immunosuppressive agents within 7 days prior to apheresis, except for the following: use of topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; short-term use of corticosteroids for prophylactic purposes (e.g., prevention of contrast agent allergy).
* 16.Administration of live attenuated vaccines within 4 weeks prior to apheresis.
* 17.Major surgery within 2 weeks prior to apheresis, or planned surgery during the study period (Note: Study participants scheduled for local anesthesia surgery may participate in this study).
* 18.History of severe allergic reactions, or hypersensitivity to any drugs or related excipients specified in the protocol, as determined by the investigator to be unsuitable for enrollment.
* 19.Any condition that, in the opinion of the investigator, makes the study participant unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-28 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Within 28 days of CG-102-12C infusion
  Describe the adverse events of limiting further increases in the dose of CG-102-12C
Treatment-emergent adverse events (TEAEs) | Within 24 months after the treatment
  Describe adverse events (AEs) and serious adverse events (SAEs) that are related to the study treatment during the treatment period.

SECONDARY OUTCOMES:
Objective response rate (ORR) | From treatment of the first subject to completion of follow-up of the last subject (up to 5 years)
  Objective response rate by RECIST 1.1.
Disease control rate (DCR) | within 1 year after the last subject was treated
  The proportion of patients whose disease is controlled, which includes those who achieve a complete response (CR), partial response (PR), or stable disease (SD), out of the total number of evaluable patients.
Duration of remission (DOR) | From enrollment of the first subject to completion of follow-up of the last subject (up to 5 years)
  Duration of response by RECIST 1.1
Time to remission (TTR) | From enrollment of the first subject to completion of follow-up of the last subject (up to 3 years)
  Time to remission by RECIST 1.1
Progression free survival (PFS) | From enrollment of the first subject to completion of follow-up of the last subject (up to 5 years)
  Progression-free survival by RECIST 1.1
Overall survival (OS) | From enrollment of the first subject to completion of follow-up of the last subject (up to 5 years)
  Overall survival by RECIST 1.1.
CAR-T Cmax | Within 28 days of CG-102-12C infusion
  Describe the peak concentration of CG-102-12C in vivo
CAR-T Tmax | Within 28 days of CG-102-12C infusion
  Describe the time from infusion to reaching peak concentration of CG-102-12C in vivo

OTHER OUTCOMES:
Immune cell subsets endpoint | Within 28 days of CG-102-12C infusion
  The proportion of peripheral blood immune cells at different sampling points before and after the reinfusion of CG-102-12C injection.
Cytokine / inflammation related protein endpoint | Within 28 days of CG-102-12C infusion
  IL-2, IL-2 and IL-2 before and after reinfusion of CG-102-12C injection The concentration levels of IL-6, IL-15, IL-21, IFN-γ, TNF α, C-reactive protein, ferritin.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - First Affiliated Hospital, Medical College of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No